CLINICAL TRIAL: NCT06448559
Title: Feedback From Patients, Informal Caregivers and Healthcare Professionals on the New Profession of Care Manager in Maintenance Pulmonary Rehabilitation Programmes: a Qualitative Study
Brief Title: Feedback on the New Profession of Care Manager in Maintenance Pulmonary Rehabilitation Programmes
Acronym: RECOORDS
Status: Completed | Type: Observational
Sponsor: GCS CIPS (Other)
Responsible Party: Sponsor
Other Study IDs: RECOORDS
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with Chronic obstructive pulmonary disease (COPD): Patients who have joined a long-term and remote Maintenance Pulmonary Rehabilitation Programmes (M-PRP) No intervention Semi-directive interview
  Interventions: Other: Semi-directive interview
- Informal caregivers: Informal caregivers designated by patients who participated in M-PRP No intervention Semi-directive interview
  Interventions: Other: Semi-directive interview
- Care-managers: Health professionals who have carried out the mission of monitoring coordinator (care-manager) within the framework of a M-PRP No intervention Semi-directive interview
  Interventions: Other: Semi-directive interview

INTERVENTIONS:
Other: Semi-directive interview — Semi-directive interviews are individual interviews used in a qualitative approach to collect information in order to perform a thematic analysis

SUMMARY:
Pulmonary rehabilitation (PR) is one of the main treatments for COPD, but its benefits are transient. The care manager's mission is to help the patient maintain the long-term benefits of their stay by adopting health-promoting behaviors and anticipating the risks of dropping out. To do this, it has IT tools allowing it to monitor the patient remotely. He/She remains in contact with the patient and discussion times are regularly scheduled; It also relies on the multidisciplinary team of the PR center to guide the patient when needs are identified.

As the experiments have not yet been completed, the effectiveness and efficiency data (cost-economic ratio) are not yet known. However, beyond these highly anticipated quantitative results, these experiments do not plan to analyze this new mode of support on a qualitative side. Even if they prove favorable, the quantitative results will in no way predict the success of the deployment of this type of support on a large scale. Taking into account the opinions of users, but also the difficulties encountered or potential points of improvement are all important data to take into account in order to successfully implement this new profession outside the framework and controlled context of the experimentation. Consequently, we aim to conduct a qualitative study with feedback from patients participating in ongoing healthcare professional experiments, on the new profession of care manager. We also want to interview their informal caregivers and health professionals practicing this new profession.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) is one of the main treatments for COPD, but its benefits are transient. Indeed, patients generally return to their initial state of health within 6 months to 1 year after the PR stay. To increase long-term effectiveness, several recent studies have experimented with maintenance PR programmes (M-PRPs), orchestrated by a care manager. The care manager's mission is to help the patient maintain the long-term benefits of their stay by adopting health-promoting behaviors and anticipating the risks of dropping out. To do this, it has IT tools allowing it to monitor the patient remotely, such as a digital monitoring solution (educational sheets, shared calendar, videoconferencing tool, etc.) and connected objects (scales, blood pressure monitor, etc.). He/She remains in contact with the patient and discussion times are regularly scheduled (once or several times per month). It also relies on the multidisciplinary team of the PR center to guide the patient when needs are identified.

This mode of support based on the emergence of a new profession seems promising because it responds to a real need shared by patients, namely the need to be supported beyond the temporary bubble of the PR stay, while relying on telecommunications tools in order to be part of an economically reasoned approach. As the experiments have not yet been completed, the effectiveness and efficiency data (cost-economic ratio) are not yet known. However, beyond these highly anticipated quantitative results, these experiments do not plan to analyze this new mode of support on a qualitative side. However, even if they prove favorable, the quantitative results will in no way predict the success of the deployment of this type of support on a large scale. Taking into account the opinions of users, but also the difficulties encountered or potential points of improvement are all important data to take into account in order to successfully implement this new profession outside the framework and controlled context of the experimentation. Thus, we wish to conduct a qualitative study with feedback from patients participating in ongoing healthcare professional experiments, on the new profession of care manager. We also want to interview their informal caregivers and health professionals practicing this new profession.

ELIGIBILITY:
Inclusion Criteria:

1. For COPD patients

   * Patients who have joined a long-term and remote M-PRP.
   * Patients followed or having been followed for more than 6 months by a care manager
   * Patients who have attended at least 30% of follow-up interviews
2. For Informal Caregivers

   * Informal caregivers designated by patients who participated in M-PRP
   * A person who meets the definition of a carer under article L.113-1-3 of the law of 28/12/2015 relating to the adaptation of society to ageing (www.legifrance.gouv.fr/loda/article_lc/JORFARTI000031701024/) i.e.: 'The following are considered to be close carers of an elderly person: their spouse, the partner with whom they have entered into a civil solidarity pact or their cohabitee, a parent or an ally, defined as family carers, or a person living with them or maintaining close and stable ties with them, who helps them, on a regular and frequent basis, on a non-professional basis, to carry out all or part of the acts or activities of daily life.'
   * Person meeting the criteria of carer for more than 6 months
3. For Care-managers

   * Health professionals who have carried out the mission of care-manager within the framework of a M-PRP
   * Health professional who is or has been a care-manager for more than 6 months
   * Care-manager who follows or has followed more than 10 patients

Exclusion Criteria:

1. For COPD patients

   * Protected adults, vulnerable persons
   * Patients who completed their M-PRP more than 4 months ago.
2. For Informal Caregivers

   * Minors, protected adults, vulnerable persons
   * Helped patients who have completed their M-PRP for more than 4 months.
3. For Care-managers

   * No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients, informal caregivers and care-managers participating in a M-PRP
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Typology and categorization of definition and perception of the profession of care manager | During M-PRP or just after completion
  collected through interviews with each group
Typology and categorization of technical aspect / modalities of the profession of care-manager | During M-PRP or just after completion
  collected through interviews with each group
Typology and categorization of areas for improvement concerning the profession of care manager | During M-PRP or just after completion
  collected through interviews with each group

CONTACTS AND LOCATIONS:
Overall Officials: Nelly HERAUD, PhD, Study Director — CLARIANE
Locations (1):
- Clinique Souffle La Vallonie, Lodève, France

IPD SHARING:
Plan to Share IPD: Undecided